CLINICAL TRIAL: NCT02978300
Title: High-Flow Nasal Cannula Oxygen Therapy (HFNC) Alone or Associated With Noninvasive Ventilation (NIV) for Immunocompromised Patients Admitted to Intensive Care Unit for Acute Respiratory Failure : FLORALI-Immunodéprimés
Brief Title: HFNC Alone or Associated With NIV for Immunocompromised Patients Admitted to ICU for Acute Respiratory Failure
Acronym: FLORALI-IM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-A00834-47
Record Dates: First submitted 2016-11-24; First posted 2016-11-30 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Acute Respiratory Failure; Immunosuppression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NIV/HFNC group (Active Comparator): Continuous NIV for at least 4 hours until clinical improvement then intermittent 1-hour sessions for a minimal duration of 12 hours a day. Between NIV sessions HFNC will be delivered as in the HFNC group.
  Interventions: Device: NIV/HFNC
- HFNC group (Experimental): Continuous HFNC alone 24h/24 until weaning or intubation.
  Interventions: Device: HFNC

INTERVENTIONS:
Device: NIV/HFNC — Pressure support level to achieve an expired tidal volume between 6 and 8 ml/kg of predicted body weight Positive end expiratory pressure from 5 to 10 cm H2O, aiming a PEEP level ≥ 8 cm H2O FiO2 set to achieve SpO2 ≥ 92%
  Arms: NIV/HFNC group
Device: HFNC — Gas flow of 60 l/min and FiO2 set to achieve SpO2 ≥ 92%
  Arms: HFNC group

SUMMARY:
Acute respiratory failure is the leading cause of ICU admission of immunocompromized patients. In this subgroup of patients, the need for intubation and invasive mechanical ventilation occurs in about 50% of cases and is associated with very a high mortality rate, reaching 70% of cases. Therefore, noninvasive oxygenation strategies have been developed to avoid intubation.

More than 15 years ago, 2 trials have suggested that NIV could decrease intubation and mortality rates of immunocompromized patients as compared to standard oxygen through a mask. However these results have not been confirmed in a recent large trial.

HFNC is a recent and well-tolerated oxygenation technique. In a recent trial, HFNC alone could decrease mortality and intubation rates in patients with ARF as compared to NIV. Similar findings have been reported in a post-hoc analysis on immunocompromized patients excluding those with profound neutropenia. Likewise in a retrospective monocentric cohort of immunocompromized patients, we reported better outcomes with HFNC than with NIV.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Admission to ICU for acute respiratory failure defined by all of the following criteria:

  * Dyspnea at rest with RR ≥ 25 breaths/min
  * PaCO2 ≤ 50 mm Hg
  * PaO2/FiO2 ≤ 300 mm Hg under oxygen ≥ 10 l/min through a mask or HFNC or NIV (for patients under oxygen FiO2 will be calculated using the following formula: oxygen flow in liters per minute x 3 + 21)
* Immunosuppresion defined by 1 of the following criteria:

  * Hematological malignancy (active or remitting < 5 years)
  * Allogenic stem cell transplantation < 5 years
  * Solid cancer (active)
  * Leucopenia < 1 G/l or neutropenia ≤ 0.5 G/l after chemotherapy
  * Solid organ transplantation
  * AIDS (not only HIV)
  * Treatment with immunosuppressive or immunomodulatory drugs
  * Systemic steroids ≥ 0.5 mg/kg/d of prednisone-equivalent for ≥ 3 weeks
* Non opposition to participate obtained from the patient or their legally acceptable representative.

Exclusion Criteria:

* Contraindication of NIV (patient refusal, cardiac arrest, coma, not drained pneumothorax, unresolving vomiting, upper airways obstruction, hematemesis, severe facial trauma)
* Chronic respiratory failure with altered pulmonary function tests
* Overt cardiogenic pulmonary edema
* Urgent need for intubation
* Severe shock (vasopressors > 0.3 µg/kg/min to maintain SAP > 90 mm Hg)
* Impaired consciousness (Glasgow coma scale score ≤ 12) or agitation
* Surgery under general anesthesia < 7 days
* Previously included in the trial
* Do-not-intubate order
* Pregnancy or breastfeeding
* Persons benefiting from enhanced protection, namely minors, persons deprived of their liberty by a judicial or administrative decision, persons staying in a health or social institution, adults under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2017-01-21 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
mortality rates | day 28
  Mortality rates at day 28 after randomization will be compared between the 2 groups

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Coudroy, M.D., Study Director — Poitiers University Hospital
Locations (1):
- CHU de Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Coudroy R, Frat JP, Ehrmann S, Pene F, Terzi N, Decavele M, Prat G, Garret C, Contou D, Bourenne J, Gacouin A, Girault C, Dellamonica J, Malacrino D, Labro G, Quenot JP, Herbland A, Jochmans S, Devaquet J, Benzekri D, Vivier E, Nseir S, Colin G, Thevenin D, Grasselli G, Assefi M, Guerin C, Bougon D, Lherm T, Kouatchet A, Ragot S, Thille AW; REVA Network. High-flow nasal oxygen therapy alone or with non-invasive ventilation in immunocompromised patients admitted to ICU for acute hypoxemic respiratory failure: the randomised multicentre controlled FLORALI-IM protocol. BMJ Open. 2019 Aug 10;9(8):e029798. doi: 10.1136/bmjopen-2019-029798. PMID 31401603
- [Derived] Coudroy R, Frat JP, Ehrmann S, Pene F, Decavele M, Terzi N, Prat G, Garret C, Contou D, Gacouin A, Bourenne J, Girault C, Vinsonneau C, Dellamonica J, Labro G, Jochmans S, Herbland A, Quenot JP, Devaquet J, Benzekri D, Vivier E, Nseir S, Colin G, Thevenin D, Grasselli G, Bougon D, Assefi M, Guerin C, Lherm T, Kouatchet A, Ragot S, Thille AW; FLORALI-IM study group and the REVA Research Network. High-flow nasal oxygen alone or alternating with non-invasive ventilation in critically ill immunocompromised patients with acute respiratory failure: a randomised controlled trial. Lancet Respir Med. 2022 Jul;10(7):641-649. doi: 10.1016/S2213-2600(22)00096-0. Epub 2022 Mar 21. PMID 35325620